CLINICAL TRIAL: NCT04078646
Title: Influence of Proteins on the Bioavailability of Carotenoids
Acronym: CAROPROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Laboratoires Réunis (Unknown); Université Catholique de Louvain (Other); Luxembourg Institute of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 201710/04
Record Dates: First submitted 2019-08-08; First posted 2019-09-06 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Absorption; Chemicals; Healthy Diet; Metabolism
Keywords: Carotenoids; Postprandial absorption; Area-under-curve; Bioavailability; Proteins; Tomato juice; Carrot juice; Randomized cross-over
MeSH Terms: interventions — Methods; Soybean Proteins; Whey Proteins

STUDY DESIGN:
Intervention Model Description: Twenty four male individuals from or living in the region of Luxembourg will be recruited for this study. The number of participants is based on a randomized block design, constituting of 6 blocks of 4 subjects, each will be served different sequences of test meals (A, B, C/A, C, B/B, C, A/B, A, C/C, A, B/C, B, A) in order to cancel out any potential effect of sequence of meals.
  Thus, each subject will act has his/her own control. Test meal intake will be separated by 1 week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary intervention (Experimental): Intervention with test meal only
  Interventions: Other: Intervention without protein addition
- Dietary intervention 2 (Experimental): Intervention with test meal and whey protein isolate (30 g)
  Interventions: Other: Intervention with whey protein
- Dietary intervention 3 (Experimental): Intervention with test meal and soy protein (30 g)
  Interventions: Other: Intervention with soy protein isolate

INTERVENTIONS:
Other: Intervention with soy protein isolate — Test meals will be served to the subjects, containing soy protein isolate:
  350 mL carrot/tomato juice (50:50, v/v), with 30 g added soy protein, plus 5 ml peanut oil
  as morning test meal, served together with 40 g toasted bread and 20 g of cream-cheese plus 10 g margarine.
  Arms: Dietary intervention 3
Other: Intervention with whey protein — Test meals will be served to the subjects, containing soy protein isolate:
  350 mL carrot/tomato juice (50:50, v/v), with 30 g added whey protein isolate, plus 5 ml peanut oil
  as morning test meal, served together with 40 g toasted bread and 20 g of cream-cheese plus 10 g margarine.
  Arms: Dietary intervention 2
Other: Intervention without protein addition — Test meals will be served to the subjects, containing soy protein isolate:
  350 mL carrot/tomato juice (50:50, v/v), plus 5 ml peanut oil
  as morning test meal, served together with 40 g toasted bread and 20 g of cream-cheese plus 10 g margarine.
  Arms: Dietary intervention

SUMMARY:
A postprandial intervention study is conducted on healthy male subjects to evaluate whether the addition of proteins (why protein isolate, soy protein) can help to increase the bioavailability of carotenoids from a tomato/carrot beverage.

DETAILED DESCRIPTION:
Participants who agree to sign the Informed Consent Form and are considered eligible for participation will be scheduled for a first and brief screening visit enrolment visit) to collect a spot urine and blood sample (20 ml) that are meant to check the subjects anemic status and analyze the sugar levels as well as plasma lipids such as triglycerides, in order to screen for any abnormal health condition (e.g. onset of diabetes) that they might not be aware of at the date of the information session and that might not make them eligible for this study.

If at this stage they are still considered eligible for the study, participants will commence the 4 week trial phase which includes 3 washout periods, 1 short screening visit and 3 full day (i.e. 10.5 hours) clinical visits. The screening visit, called preliminary visit, will take place at the beginning of the trial phase. A blood sample will be collected to determine the baseline levels of triglycerides and plasma carotenoids at the beginning of the trial, prior to the first washout phase.

The first washout week starts on day 1 after the preliminary visit and will have a duration of 14 days during which the participants will be asked to stay on a low carotenoid diet (i.e. to avoid the intake of colored fruits and vegetables), to reduce the basal levels of blood circulating carotenoids.

During the 1-day appointments at the Clinical and Epidemiological Investigation Centre (CIEC), one of the three test meals will be given to the participants in 6 different orders, making 6 treatment patterns. Assuming that all 24 participants are successfully recruited, we will have 4 randomly allocated participants per pattern.

On clinical visit days, participants will be asked to report at the CIEC's facilities, starting from 7:30 am, and a baseline blood sample (20 ml) will be drawn at 0h time point. A trained nurse will insert a cannula in the forearm of the participant that will be left in place during the whole staying for the commodity of the participant.

Immediately after the baseline blood draw, a test meal composed of a mixture of carrot and tomato juice (350 mL in total), to which 5 mL of peanut oil will be added, 40 g of toasted bread (white wheat, with 10 g margarine plus 20 g cream-cheese) and a glass of water (approx. 300 mL) which may or may not contain 30 g of proteins (either a plant based protein or a dairy-based proteins) will be served. The entire test meal must be eaten within 30 min, under supervision.

Post-prandial blood samples (20 ml each) will be collected at timed intervals (before, 2h, 3h, 4h, 5h. 6h, 8h and 10h after test meal intake). Participants will receive a standardized lunch 4 hours after test meal intake (c.a. 12:00 pm), consisting of a toasted sandwich (white wheat bread, ca 60 g), with ca. 60 g turkey with some margarine to spread on the bread (ca 10 g), a Greek yogurt (140 g) and a small apple. A courtesy meal 10 hours after test meal intake for dinner and at the end of the visit. No other foods or beverages except water (ad libitum) will be allowed during the day (including during breakfast and lunch if desired).

This first clinical appointment will be followed by a 1 week washout period, during which he/she will continue on a low carotenoid diet (3rd week of washout diet). At the end of the 3rd week of washout, the second appointment at the LIH clinical center will take place. The procedure for this day is the same as mentioned above. The second appointment is followed by the 4th and last washout week and at the end the participant will have the 3rd and last appointment at the Luxembourg Institute of Health (LIH) clinical center, which will be identical to the other visits. For all washout periods the participants will be asked to fill a provided food journal, on a daily basis, where they will write down what they have eaten during the day. This will be used to check compliance with the washout period and better interpret personal data.

Stool collection: For a limited number of subjects (n=6), the samples will be collected following intake of all 3 test meals. For this purpose, Containers for collection and plastic clip-bags and bags will be handed to participants. Boxes with cooling elements for stool collection will likewise be given. Also, six fecal color markers will be provided to the participants. For each clinical visit, two fecal marker are needed. Collections will start from the excretion of the first fecal color marker (brilliant blue) which will be taken at the beginning of the fasting period, i.e. the day before each clinical day. The collection will continue to the excretion of the second fecal marker which should be taken on the morning of the day following each clinical visit (before breakfast). Samples will be returned after the clinical test day as soon as the last fecal marker has been excreted (normally resulting in 2-3 day complete fecal samples), and could be collected once in between by staff from the LIH if needed.

ELIGIBILITY:
Inclusion Criteria:

* healthy and free living;
* men;
* age between 20 and 50 years old;
* Body-Mass-Index (BMI) <30 kg/m2
* non-smokers (abstinent for more than 2 years);

Exclusion Criteria:

* suffering from any metabolic disease that may cause digestive disturbances (such as Crohn's disease or colitis);
* malabsorption disorders;
* BMI over 30 kg/m2;
* hyperlipidaemia (triglycerides and total cholesterol over 200 mg/dl)
* any individuals following a special diet that is not compatible with wash-out periods or test meals (vegetarian, gluten-free or diabetic);
* regular consumption of more than 5 portions (80-100 g) of fruits and vegetables per day;
* being on medical treatment or consuming any medication for chronic conditions or recent illness (e.g. antibiotics);
* consuming regularly dietary supplements;
* abnormally high or low values of plasma circulating carotenoids;
* tobacco smoking;
* frequent alcohol consumption (over 2 glasses per day);
* food allergies or intolerances that are not compatible with test meals (e.g. gluten or milk intolerance);
* daily practice of intense physical activity of 120 min or more.

No special population group such as prisoners, children, the mentally disabled or groups whose ability to give voluntary informed consent may be in question, will be recruited for this study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only self-declared men will participate in the study
Enrollment: 24 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Concentration of carotenoids in plasma triacyl-rich-lipoprotein (TRL) fraction | 10 hours postprandial, measured on 3 test clinical test days after test meal intake, interspersed by 1 week each
  Carotenoid concentration (lycopene, beta-carotene) studied over 10 hours postprandial (area-under curve of concentration vs. time)

SECONDARY OUTCOMES:
Time of maximum concentration of lycopene and beta-carotene and triglycerides in plasma-TRL fraction | 10 hours postprandial, measured on 3 clinical test days after test meal intake, interspersed by 1 week
  Studying the timely appearance of carotenoids in the plasma TRL fraction, i.e. the time when concentration with reach a maximum
Maximum concentration of lycopene and beta-carotene and triglycerides in plasma-TRL fraction | 10 hours postprandial, measured on 3 test clinical days after test meal intake, interspersed by 1 week
  Studying the maximum concentration of lycopene and beta-carotene in the plasma-TRL fraction, i.e. the maximum concentration reached during the 10 h monitoring
Fecal degradation products of carotenoids | Collection covering the test meal intake period, starting from the excretion of a brilliant blue capsule taken the 12 hours before test meal intake, until complete excretion of a second brilliant blue capsule taken 24 hours after test meal intake
  Studying native carotenoids and degradation products in pooled stool excreted following test meal intake (fecal balance method), i.e. the stool collected following test meal intake

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Bohn, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No
Data of subjects will not be available for outside researchers.

REFERENCES:
- [Background] Iddir M, Degerli C, Dingeo G, Desmarchelier C, Schleeh T, Borel P, Larondelle Y, Bohn T. Whey protein isolate modulates beta-carotene bioaccessibility depending on gastro-intestinal digestion conditions. Food Chem. 2019 Sep 1;291:157-166. doi: 10.1016/j.foodchem.2019.04.003. Epub 2019 Apr 1. PMID 31006454
- [Background] Soukoulis C, Bohn T. A comprehensive overview on the micro- and nano-technological encapsulation advances for enhancing the chemical stability and bioavailability of carotenoids. Crit Rev Food Sci Nutr. 2018 Jan 2;58(1):1-36. doi: 10.1080/10408398.2014.971353. Epub 2017 Jul 5. PMID 26065668
- [Result] Corte-Real J, Guignard C, Gantenbein M, Weber B, Burgard K, Hoffmann L, Richling E, Bohn T. No influence of supplemental dietary calcium intake on the bioavailability of spinach carotenoids in humans. Br J Nutr. 2017 Jun;117(11):1560-1569. doi: 10.1017/S0007114517001532. Epub 2017 Jun 27. PMID 28651681
- See also: Description of study — https://www.luxclin.lu/Articles/Details/?c=ART0312NUJ
- See also: Funding information — https://www.fnr.lu/core-2016-call-funding-results/

DOCUMENTS (3):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04078646/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04078646/SAP_000.pdf
  • Informed Consent Form (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04078646/ICF_001.pdf